CLINICAL TRIAL: NCT00484991
Title: Sapropterin Expanded Access Program
Status: Approved for marketing | Type: Expanded Access
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: BioMarin BPPS, BioMarin Pharmaceutical Inc.
Other Study IDs: SEAP-001
Record Dates: First submitted 2007-06-08; First posted 2007-06-12 (Estimated); Last update posted 2008-04-15 (Estimated); Status verified 2008-04

CONDITIONS: Phenylketonuria
Keywords: Phenylketonuria; PKU; Phenylketonurias; Hyperphenylalaninaemia; Hydroxylase Deficiency
MeSH Terms: conditions — Phenylketonurias | interventions — sapropterin; phenoptin

INTERVENTIONS:
Drug: Sapropterin dihydrochloride — 20mg/kg/day orally, physicians may adjust the dose within a range of 5-20mg/kg/day as warranted by their clinical judgment.
  Other Names: Kuvan; Phenoptin

SUMMARY:
The Purpose of this study is to provide patients with hyperphenylalaninemia (HPA) due to Phenylketonuria (PKU) access to sapropterin dihydrochloride and to collect more information about the safety of the drug in an expanded access program (EAP) until commercial product is available.

DETAILED DESCRIPTION:
The sapropterin EAP (SEAP) is an open-label, multi-center program designed to provide access to sapropterin dihydrochloride for patients diagnosed with hyperphenylalaninemia due to PKU. All patients with a confirmed diagnosis of hyperphenylalaninemia due to PKU who are not currently enrolled in a clinical study with sapropterin dihydrochloride and meet the requisite inclusion criteria and do not meet any of the exclusion criteria may be eligible to participate in this program. Eligible patients may receive sapropterin dihydrochloride and participate in the program until commercial drug is available, however, the program will not continue beyond 2 months after the product receives marketing approval from the FDA. During the program, physicians will use their clinical judgment to assess whether a patient is a responder to sapropterin dihydrochloride. Participating physicians will measure blood Phe levels at baseline prior to treatment and then at least once between Day 7 and Day 30 following initiation of treatment to determine if the patient is a responder. A responder is a patient that has a clinically significant reduction in either the absolute or percent decrease in blood phenylalanine level compared to pre-treatment levels. The recommended starting dose of sapropterin dihydrochloride is 20 mg/kg/day. Physicians treating their patients with sapropterin dihydrochloride will be able to adjust the dose within a range of 5 mg/kg/day to 20 mg/kg/day if warranted in their clinical judgment. Adverse event information will be collected in an ongoing fashion through patient reporting AEs to their physician. Physicians will ask patients for information regarding adverse events that have occurred since the last visit. An adverse event report form will be completed in these cases and sent to BioMarin.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has hyperphenylalaninemia due to PKU, a rare and serious disease
2. Patient is not participating in a sapropterin dihydrochloride clinical study
3. Patient is older than 8 years of age
4. Patient is willing and able to provide written informed consent or, in the case of under the age of 18, provide written assent (if required) and written informed consent by a parent or legal guardian
5. If female and of child bearing potential, the patient has a negative urine pregnancy test within 24 hours prior to enrollment (females of child-bearing potential only) and will be using adequate contraceptive methods to avoid pregnancy while participating in the program
6. Patient is willing and able to comply with program procedures
7. Patient lives in the United States

Exclusion Criteria:

1. Patient is perceived to be unreliable or unwilling to comply with program participation or, if under the age of 18, have parents or legal guardians who are perceived to be unreliable or unwilling to comply with program participation
2. Patient has a concurrent disease or condition that would interfere with program participation or safety
3. Patient is 8 years old or younger
4. Patients is eligible for enrolling in PKU-010
5. Patient is participating in an ongoing study with sapropterin dihydrochloride
6. Patient is pregnant, breast feeding or considering pregnancy
7. Patient is taking levodopa

Min Age: 9 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (36):
- United States (36):
  - Los Angeles, California
  - Orange, California
  - San Diego, California
  - Stanford, California
  - Denver, Colorado
  - Gainseville, Florida
  - Tampa, Florida
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Bangor, Maine
  - Boston, Massachusetts
  - Minneapolis, Minnesota
  - Columbia, Missouri
  - Kansas City, Missouri
  - St Louis, Missouri
  - Newark, New Jersey
  - Manhasset, New York
  - Rochester, New York
  - Stony Brook, New York
  - Valhalla, New York
  - Akron, Ohio
  - Columbus, Ohio
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Florence, South Carolina
  - Sioux Falls, South Dakota
  - Galveston, Texas
  - Houston, Texas
  - Salt Lake City, Utah
  - Charlottesville, Virginia
  - Norfolk, Virginia
  - Madison, Wisconsin
  - Milwakee, Wisconsin